CLINICAL TRIAL: NCT03427879
Title: Effect of Flavonoids on Gut Permeability in Cyclists
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Utah State University (Other)
Responsible Party: Principal Investigator, Robert Ward, Associate Professor, Utah State University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 1010820
Record Dates: First submitted 2018-01-30; First posted 2018-02-09 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Gut Permeability, Gut Inflammation

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low flavonoid beverage (Placebo Comparator): Subjects will consume 310 milliliters per day of a dairy-based, low flavonoid, sports nutrition recovery beverage 14 days.
  Interventions: Drug: Low flavonoid beverage
- High flavonoid beverage (Active Comparator): Subjects will consume 310 milliliters per day of a dairy-based, high flavonoid, sports nutrition recovery beverage 14 days.
  Interventions: Drug: High flavonoid beverage

INTERVENTIONS:
Drug: Low flavonoid beverage — A low flavonoid, sports nutrition recovery beverage will be prepared from milk (78%), sugar (8.6%), maltodextrin (8.6%), placebo blueberry powder (2.4%), alkalized cocoa powder (1.6%), and whey protein isolate (0.6%). The beverage will contain approximately 5mg flavonoids per serving.
  Arms: Low flavonoid beverage
Drug: High flavonoid beverage — A high flavonoid, sports nutrition recovery beverage will be prepared from milk (78%), sugar (8.6%), maltodextrin (8.6%), blueberry powder (2.4%), cocoa powder (1.6%), green tea extract (0.1%) and whey protein isolate (0.6%). The beverage will contain approximately 620 mg flavonoids per serving.
  Arms: High flavonoid beverage

SUMMARY:
The purpose of this investigation is to test the hypothesis that chronic supplementation with a dairy-based beverage containing a mixture of blueberry, green tea, and cocoa flavonoids (non-nutritive natural plant compounds) will ameliorate exercise-related changes in gut permeability and inflammation. In a previous feeding study in humans, (NCT02728570) a high flavonoid diet (flavonoids at 340 mg/1000kcal) was effective in mitigating gut permeability and inflammation in overweight and obese adults compared to a low flavonoid diet (10mg/1000 kcal). To test this hypothesis, 20 trained cyclists will complete a randomized crossover study with supplementation for 2 weeks with a dairy-based sports beverage containing either a high flavonoid (approximately 620 mg) or low flavonoid (approximately 5mg) beverage. After the two week intervention, cyclists will complete a 1 hour cycling trial (45 min at 65% VO2 max then 15 minute time trial). The primary endpoints will be gut permeability as measured by plasma intestinal fatty acid binding protein (I-FABP) and the differential sugar test. Secondary endpoints will include gut inflammation (measured via fecal calprotectin), plasma cytokines (IL-6, IL-10 and TNFα) and plasma LPS. In addition, the distance completed in the time trial is a secondary endpoint.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of any race or ethnicity between 18 to 49 years of age
* Competed in a road race or triathlon in past 12 months
* Free of chronic disease and GI conditions
* Train at least 3 times per week, 1 hour at a time on average
* Willing to prepare and consume provided pre-workout beverage daily
* Maintain weight (no more/less than 5 kg change)
* Willing to avoid consumption of high flavonoid foods/supplements, large dose vitamin and mineral supplements, and NSAIDs or other medications known to affect inflammation during study period
* Willing to provide urine, stool, and blood samples

Exclusion Criteria:

* Age <18 or >50 years
* Medical history of heart disease, hypertension, diabetes, Crohn's disease, IBS, colitis, celiac disease, inflammatory or autoimmune disease, and lactose intolerance
* Uncontrolled hypertension: diastolic blood pressure >95 mm Hg or systolic blood pressure >160 mm Hg
* For women: pregnancy, breast feeding or postpartum <6 months
* Food allergies or restrictions to treatment/placebo beverages
* Chronic use of NSAIDs
* Consumption of flavonoid supplements <1 month prior to study start
* Antibiotic use <3 months prior to study start
* Other conditions (medical, psychiatric, or behavioral) that may present a safety hazard to the participant or interfere with study participation, as determined by the principal investigators

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-09-14 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-07-31 (Actual)

PRIMARY OUTCOMES:
Urinary lactulose:mannitol ratio by gas chromatography | Three weeks
  Measure of gut permeability from mouth to end of small intestine. Ratio of urinary lactulose to mannitol after subject consumes a beverage containing these sugars. Sugars in urine are measured by gas chromatography with flame ionization detection.
Plasma intestinal fatty acid binding protein (i-FABP) by ELISA | Three weeks
  Marker of gut wall integrity. i-FABP is measure by enzyme-linked immunosorbent assay in plasma of subjects after the time trial.

SECONDARY OUTCOMES:
Fecal calprotectin by ELISA | Three weeks
  Secondary endpoint for intestinal inflammation. Calprotectin is measured in fecal samples by enzyme-linked immunosorbent assay.
Urinary sucralose:mannitol ratio by gas chromatography | Three weeks
  Secondary measure of gut permeability from mouth to end of colon. Ratio of urinary lactulose to mannitol after subject consumes a beverage containing these sugars. Sugars in urine are measured by gas chromatography with flame ionization detection.
Serum soluble tumor necrosis factor (TNFa) by ELISA | Three weeks
  One of four secondary endpoints for systemic inflammation. The cytokine, TNFa, is measured in plasma by enzyme-linked immunosorbent assay.
Serum soluble interleukin-6 (IL-6) by ELISA | Three weeks
  One of four secondary endpoints for systemic inflammation. The cytokine, IL-6, is measured in plasma by enzyme-linked immunosorbent assay.
Serum soluble interleukin-10 by ELISA | Three weeks
  One of four secondary endpoints for systemic inflammation. The cytokine, IL-10, is measured in plasma by enzyme-linked immunosorbent assay.
Serum endotoxin by ELISA. | Three weeks
  One of four secondary endpoint for systemic inflammation. The bacterial cell wall product is measured in plasma by enzyme-linked immunosorbent assay.
Distance ridden in time trial | One Day
  Subjects will complete a 15m time trial on a bike after each dietary intervention. The distance covered in each time trial will be measured by the computer on the exercise bike.
Rating of perceived exertion by questionnaire. | One Day
  Subjects will complete a 15m time trial on a bike after each dietary intervention. This measure is a subjective measure of the difficulty of the work. Subjects will provide the ratings orally during the time trial.

CONTACTS AND LOCATIONS:
Overall Officials: Robert E Ward, PhD, Principal Investigator — Nutrition, Dietetics and Food Sciences, Utah State University
Locations (1):
- Center for Human Nutrition Studies, Logan, Utah, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kung S, Vakula MN, Kim Y, England DL, Bergeson J, Bressel E, Lefevre M, Ward R. No effect of a dairy-based, high flavonoid pre-workout beverage on exercise-induced intestinal injury, permeability, and inflammation in recreational cyclists: A randomized controlled crossover trial. PLoS One. 2022 Nov 29;17(11):e0277453. doi: 10.1371/journal.pone.0277453. eCollection 2022. PMID 36445874